CLINICAL TRIAL: NCT05434936
Title: Ovarian Tissue Cryopreservation for Fertility Preservation in Girls and Women Facing a Fertility Threatening Medical Diagnosis or Treatment Regimen
Brief Title: Ovarian Tissue Cryopreservation for Fertility Preservation in Girls and Women
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Temporary protocol lapse
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Terri Lynn Woodard, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-40808
Record Dates: First submitted 2017-10-20; First posted 2022-06-28 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Fertility Preservation
Keywords: oncofertility
MeSH Terms: interventions — Ovariectomy

STUDY DESIGN:
Intervention Model Description: This is a tissue bank protocol in which prospectively collected specimens of ovarian tissue and a sample of whole blood will be obtained from patients who elective to cryopreserve ovarian tissue to preserve fertility. The portion of tissue designated for patient use will be cryopreserved using the slow freeze method while the portion designated for research purposed will be divided and cryopreserved using the slow freeze versus vitrification methods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Collection (Other): There is only one arm of the study, all patients enrolled will have surgery in which the attempt will be made to collect ovarian tissue.
  Interventions: Procedure: Oophorectomy

INTERVENTIONS:
Procedure: Oophorectomy — Patients undergoing surgery for any indicated procedure for fertility-threatening treatment will have attempt at collecting ovarian tissue at time of surgery.

SUMMARY:
This study will compare efficacy of ovarian tissue freezing using slow-freeze versus vitrification methods.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the efficacy of ovarian tissue cryopreservation using slow-freeze and vitrification methods in enabling long-term preservation of ovarian function and fertility, in females undergoing treatment that may cause infertility. This study will provide study participants with their own tissue to cryopreserve and reserve for future use and:

* Determine the efficacy of ovarian cryopreservation techniques.
* Provide long-term follow up for patients who have undergone ovarian tissue cryopreservation for participants' own use.

In addition to providing study participants with the future opportunity to use their tissue with the intent to reinstate ovarian function, this study will provide research tissue to the embryology research lab at the Family Fertility Center at Texas Children's Hospital that will be used to:

* Optimize techniques for ovarian tissue cryopreservation of ovarian tissue for use in future retransplantation).
* Investigate factors affecting successful maturation and quality of immature oocytes obtained from ovarian tissue including growth factors, hormones and other culture conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Female Patients only
2. 0-42 years of age.
3. Will undergo surgery, chemotherapy, drug treatment and/or radiation for the treatment or prevention of a medical condition or malignancy that places the patient at risk for impaired ovarian function and infertility OR, have a medical condition or malignancy that requires removal of all or part of one or both ovaries.
4. May have newly diagnosed or recurrent disease. Those not enrolled at the time of initial diagnosis are eligible if they have not received therapy that is viewed as likely to result in complete and permanent loss of ovarian function.
5. Signed an approved informed consent and authorization permitting the release of personal health information. The patient and/or the patient's legally authorized guardian(s) must acknowledge in writing that consent for specimen collection has been obtained, in accordance with institutional policies approved by the U.S. Department of Health and Human Services.

Exclusion Criteria:

1. Girls and women with psychological, psychiatric, or other conditions which prevent giving informed consent.
2. Girls and women whose underlying medical condition significantly increases their risk of complications from anesthesia and surgery.
3. Girls and women who are permanently menopausal, as documented by history and FSH levels.
4. Girls and women who are pregnant.

Ages: 0 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-08-11 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2027-10-10 (Estimated)

PRIMARY OUTCOMES:
Effect of vitrification and slow freeze cryopreservation methods on follicular survival | 5+ years
  Investigators will explore and compare the impact of vitrification and slow freeze cryopreservation methods by evaluating follicular survival using classic histological analysis of follicular morphology.

SECONDARY OUTCOMES:
Live birth rates in patients using cryopreserved ovarian tissue | 5+ years
  Investigators will explore reproductive outcomes of women using cryopreserved tissue by measuring the live birth rate as defined by the number of initial live births divided by the total number of ovarian tissue implantations performed.

CONTACTS AND LOCATIONS:
Overall Officials: Terri L Woodard, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital Pavilion For Women, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided